CLINICAL TRIAL: NCT01704807
Title: Duration of Spinal Manipulation Effects as Influenced by Orthotics
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LCC-12-RD0519110317
Record Dates: First submitted 2012-09-24; First posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Chronic; Orthotic Device; Applied Kinesiology; Manual Muscle Testing; Chiropractic
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention, Custom Orthotics (Active Comparator): Wearing custom foot orthotics
  Interventions: Device: foot orthotics
- Sham Foot Orthotic (Sham Comparator): Wearing sham or flat shoe insoles
  Interventions: Device: Sham foot orthotic

INTERVENTIONS:
Device: foot orthotics — Experimental wore experimental orthotics throughout the study period as much of the day as possible.
  Other Names: Foot Levelers, Full length ultra step foot orthotics
  Arms: Intervention, Custom Orthotics
Device: Sham foot orthotic — Control group wore sham insoles as much of the time as possible for the duration of the study period.
  Other Names: Foot Levelers flat insoles similar to Full Length Ultra Step
  Arms: Sham Foot Orthotic

SUMMARY:
Purpose of study: To assess the effects of wearing custom orthotics as opposed to placebo foot inserts on the duration of chiropractic correction of spinal fixations and muscle imbalances using applied kinesiology techniques.

DETAILED DESCRIPTION:
Participants with chronic lower back pain of greater than one month duration will be randomized to receive custom foot orthotics or placebo flat inserts. Both groups will receive chiropractic treatment 5 times over the course of 4 weeks following receipt of orthotics. Subjects and treating doctor will be blind to the insert type. Patients will report present, average, best and worst pain at each visit, and complete a Roland-Morris questionnaire. Secondary outcome measures will be number of fixated vertebral levels identified by motion palpation and challenge and number of muscles testing grade 4 and below from a list of 5 muscles to be tested bilaterally before and after each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Current low back pain episode present for one month or more
* No change in the past month in prescription medications affecting musculoskeletal pain
* Able to speak and understand English adequately to complete study forms
* Score on Roland-Morris questionnaire of 7.5 or higher or
* Average score on Chiropractic pain Index (Now, Average, and Worst scales from the Quadruple VAS pain scale) of 4 or higher.

Exclusion Criteria:

* Use of foot orthotics within the past 12 months
* Previous lumbar spine surgery
* Ongoing treatment for lower back pain by other health care providers other than stable prescription medications affecting musculoskeletal pain.
* Clinically significant chronic inflammatory spinal arthritis
* Severe osteoporosis for which spinal manipulation is contraindicated
* Spinal pathology or fracture
* Progressive neurologic deficits due to nerve root or spinal cord compression, including symptoms/signs of cauda equina syndrome
* History of bleeding disorder
* Known arterial aneurysm
* Pending/current litigation pertaining to back pain, including workers compensation claims
* Current pregnancy
* Lack of means of contacting which might preclude successful completion of study requirements
* Does not speak , read or understand English to an extent which would affect the subject's capacity to participate in informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Quadruple Visual Analog Pain Scale | Six weeks
  Pain present, best worst and average on a scale of 0 to 10, with 10 being the worst imaginable.
Roland-Morris Questionnaire | Six weeks
  Questionnaire listing activities of daily living, impacted by low back pain.

SECONDARY OUTCOMES:
Number of fixated vertebral levels | Six weeks
  Number of vertebral levels found to be fixated as determined by motion palpation and vertebral challenge.
Number of tested muscles grade 4 and below | Six weeks
  Number of five muscles tested bilaterally, which tested grade 4 or below in manual muscle testing.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Conable, DC, Principal Investigator — Logan College of Chiropractic/University Programs; Anthony Rosner, PhD, Principal Investigator — International College of Applied Kinesiology
Locations (1):
- Logan College of Chiropractic/University Programs, Chesterfield, Missouri, United States